CLINICAL TRIAL: NCT03101449
Title: Analysis of the Effects of Vocal Conditioning Through Semi-occluded Vocal Tract Exercises in Choir Singers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Federal University of Health Science of Porto Alegre (Other)
Responsible Party: Principal Investigator, Mauriceia Cassol, Prof. Dra. Mauriceia Cassol, Federal University of Health Science of Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 50412515.9.0000.5345
Record Dates: First submitted 2016-10-26; First posted 2017-04-05 (Actual); Last update posted 2017-04-05 (Actual); Status verified 2017-03

CONDITIONS: Voice

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group 1 (Experimental): 20 individuals of Coral UFCSPA without voice problems carry out the exercise with Finnish tube before choir practice once a week for a period of 14 weeks. The exercise will be carried out with blowing set to sound at regular frequency, with frequency variation and with the melody of "Happy Birthday"; each sequence will be held for 2 minutes with 1 minute interval between them.
  Interventions: Other: Finnish tube
- Group 2 (Experimental): 20 individuals of Coral UFCSPA without voice problems carry out the exercise straw phonation before choir practice once a week for a period of 14 weeks. The exercise will be carried out with blowing set to sound at regular frequency, with frequency variation and with the melody of "Happy Birthday"; each sequence will be held for 2 minutes with 1 minute interval between them.
  Interventions: Other: Staw phonation
- Group 3 (No Intervention): 10 individuals of Coral UFCSPA without voice problems. Untreated group.

INTERVENTIONS:
Other: Finnish tube — Practice the exercise with Finnish tube before choir practice once a week for a period of 14 weeks.
  Arms: Group 1
Other: Staw phonation — Practice the exercise straw phonation before choir practice once a week for a period of 14 weeks.
  Arms: Group 2

SUMMARY:
This research aims to evaluate the effects of vocal conditioning through two semioccluded vocal tract exercises (SOVTE) in choir singers.

DETAILED DESCRIPTION:
This research aims to evaluate the effects of vocal conditioning through two semioccluded vocal tract exercises (SOVTE) - Finnish tube and phonation in high strength straw - in vocal parameters, vocal extension profile and maximum phonation time for a period of four months in a group of singers. acoustic analysis will be performed of the average parameters of the fundamental frequency (F0), jitter, shimmer and glottal to Noise Excitation (GNE) by VoxMetria program and perceptual analysis through Consensus Assessment Perceptual Hearing the Voice Protocol (CAPE-V) three times: before the vocal conditioning, after the last meeting of the technical realization and a week after the vocal conditioning period.

ELIGIBILITY:
Inclusion Criteria:

* signing of the Informed Consent (IC).

Exclusion Criteria:

* voice disorders diagnosed by otolaryngologist physician;
* smokers;
* presence below 75% in the meetings.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-03; Primary Completion 2017-04 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Voice quality | 3 months
  Improved singing voice quality standard demonstrated by the perceptual analysis of voice with CAPE- V, in which there is a decrease in score value pre and post intervention.

SECONDARY OUTCOMES:
Mean fundamental frequency | 3 months
  Improvement of acoustic parameters, demonstrated by VoxMetria software.
Jitter | 3 months
  Improvement of acoustic parameters, demonstrated by VoxMetria software.
Shimmer | 3 months
  Improvement of acoustic parameters, demonstrated by VoxMetria software.
Glottal to Noise Excitation (GNE) | 3 months
  Improvement of acoustic parameters, demonstrated by VoxMetria software.
Profile vocal range | 3 months
  Improved profile vocal range, shown by Vocalgrama software.
Maximun phonation time | 3 months
  Improvement of maximum phonation time, demonstrated by measuring the maximum times of sustaining vowels and phonemes /s/ and /z/.

CONTACTS AND LOCATIONS:
Locations (1):
- Federal University of Health Science of Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No